CLINICAL TRIAL: NCT02142127
Title: An Open-Label, Single Oral Dose Phase I Study to Determine the Excretion Balance of Radiocarbon (i.e., the Sum of 14C-Labelled GFT505 and Its 14C-Metabolites) and to Investigate the Metabolic Profile and Pharmacokinetics of GFT505
Brief Title: Mass Balance Study of 14C-labelled GFT505 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genfit (Industry)
Collaborators: SGS Life Sciences, a division of SGS Belgium NV (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFT505-114-10; 2014-000958-10 (EudraCT Number)
Record Dates: First submitted 2014-05-16; First posted 2014-05-20 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Healthy
Keywords: GFT505; Mass balance; Pharmacokinetics; Metabolites; Healthy subjects; Healthy male volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 14C-labelled GFT505 120 mg (Experimental)
  Interventions: Drug: 14C-labelled GFT505 120 mg

INTERVENTIONS:
Drug: 14C-labelled GFT505 120 mg

SUMMARY:
Human mass-balance studies with radiolabelled study drug are needed to evaluate the amount of drug that is recovered over time via different elimination routes of the body, i.e., whole blood, blood cells, plasma, urine, feces, and expired air. The ideal case is to be able to demonstrate a (near) complete recovery (≥95 %) of the administered dose.

A good understanding of the metabolic pathway of the study drug is equally important. Mass-balance data, together with metabolic profiles in excreta, are used to characterize the biotransformation pathways of a drug and to help evaluate its drug-drug interaction potential.

To this purpose, in this study, blood, urine, and feces are collected to investigate the metabolic profile of GFT505, and plasma and urine are collected to investigate the non-radioactive pharmacokinetics of GFT505 and its principle metabolite GFT1007. Other metabolites will be investigated in plasma and urine according to the radioactivity results. Non-radioactive pharmacokinetics of GFT505 and metabolites in feces will be investigated according to the radioactivity results.

DETAILED DESCRIPTION:
This is a Phase I open-label, single oral dose and single center study of 14C-labelled GFT505 and its metabolites in healthy subjects.

After an overnight fast, subjects will be administered one dose of 14C-labelled GFT505 containing an equivalent of 120 mg of the compound with 240 mL of non-carbonated water. The total amount of administered radiocarbon will be 1.63-1.81 megaBecquerel (MBq) (44.1-48.8 μCi).

Blood, urine, and feces will be collected at scheduled time intervals from before administration of the radiolabelled study drug throughout confinement at the clinical center and thereafter, if needed. Several samples of expired carbon dioxide will be obtained up to 48 h after the administration of radiolabelled study drug.

Radiocarbon will be assayed in all available samples (whole blood, plasma, urine, feces, and expired air) by liquid scintillation spectrometry. The metabolic profile of GFT505 will be assayed in plasma, urine, and feces. Non-radioactive pharmacokinetics of GFT505 and its principle metabolite GFT1007 will be assayed in plasma and urine. Other metabolites will be investigated in plasma and urine according to the radioactivity results. Non-radioactive pharmacokinetics of GFT505 and metabolites in feces will be investigated according to the radioactivity results.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian males aged 55 to 65 years inclusive
* Body Mass Index (BMI) ≥ 18 ≤ 30 kg/m²
* Fitzpatrick skin type < 4
* No clinically relevant abnormalities in hematology and clinical chemistry parameters, blood pressure (BP) and heart rate (HR) (supine), or ECG results

Exclusion Criteria:

* History or presence of any hepatic, renal, respiratory, cardiovascular, neurologic, gastrointestinal, endocrine, immunologic, musculoskeletal, or hematologic disorder capable of altering the absorption, metabolism, or elimination of drugs, or capable of constituting a risk factor when taking the study drug, as judged by the investigator;
* Creatinine Clearance as calculated by the Cockcroft-Gault formula less than 60 mL/min;
* History of irregular bowel movements such as regular episodes of diarrhea, constipation (less than a mean of one bowel movement per day) or irritable bowel movement;
* Planning to become a father or to donate sperm within 3 months after the administration of study drug;
* History or presence of drug addiction (positive drug screen for amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, or opiates) or excessive use of alcohol (daily intake exceeding 2 units/day);
* Current use of nicotine containing products, i.e., more than 5 cigarettes or equivalent/day and the inability to stop using nicotine containing products during confinement in the clinical center;
* Large caffeine consumption (daily average of more than 6 cups of coffee or tea or more than 1L of caffeine-containing beverages) within the last year;
* Plasma levels of ALT, AST, or alkaline phosphatase (ALP) ≥1.5 x upper limit of laboratory normal range (ULN);
* Blood donation or loss of significant amount of blood within 12 weeks prior to dosing;
* Inability to understand the constraints of full urine and stool collection or inability to collect urine;
* Use of any drug treatment that could affect the outcome of the study from 14 days before the administration of the radiolabelled study drug (2 months for enzyme-inducing drugs) or 5 times the half-life of the medication, or anticipated use of concomitant therapy (except paracetamol) during the study;
* Exposure to ionizing radiations (except routine or dental radiography or radiography of the extremities), including participation in studies with radiolabelled compounds, or exposure to radioisotopes within one year prior to entry into the present study;
* Participation in another clinical study within 12 weeks prior to entry into the present study.

Ages: 55 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Excretion balance of radiocarbon in whole blood, blood cells, plasma, urine, feces, and expired air after a single oral dose of 14C-labelled GFT505. | 0-19 days
  Blood, urine, and feces will be collected at scheduled time intervals from before administration of the radiolabelled study drug throughout confinement at the clinical center and thereafter, if needed. Several samples of expired carbon dioxide will be obtained up to 48 h after the administration of radiolabelled study drug.
  Radiocarbon will be assayed in all available samples (whole blood, plasma, urine, feces, and expired air) by liquid scintillation spectrometry.

SECONDARY OUTCOMES:
Metabolic profile of GFT505 in plasma, urine, and feces. | 0- 19 days
  The metabolic profile of GFT505 will be assayed in plasma, urine, and feces. Non-radioactive pharmacokinetics of GFT505 and its principle metabolite GFT1007 will be assayed in plasma and urine. Other metabolites will be investigated in plasma and urine according to the radioactivity results. Non-radioactive pharmacokinetics of GFT505 and metabolites in feces will be investigated according to the radioactivity results.
Safety parameters | 0 - 19 days
  Safety assessment will be based on adverse events (AEs), clinical laboratory tests, electrocardiogram (ECG), vital signs, and physical examination.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Megnien, MD, Study Director — Chief Medical Officer, Genfit
Locations (1):
- SGS Life Science Services, Antwerp, Belgium